CLINICAL TRIAL: NCT02326714
Title: Effect of Auricular Acupressure on Overweight/Obese Adolescent and Young Women With Polycystic Ovary Syndrome.
Brief Title: Auricular Acupressure (AA) For Overweight/Obese Adolescent and Young Polycystic Ovary Syndrome ( PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Associate chief physician, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AA for PCOS
Record Dates: First submitted 2014-12-11; First posted 2014-12-29 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular acupressure (Experimental): The magnetic beads will be taped to the seven pressing points: Hunger point, Ovary, Uterus, Endocrine point, liver, kidney and spleen.
  Interventions: Other: Auricular acupressure
- Placebo auricular acupressure (Placebo Comparator): The magnetic beads will be taped to the three pressing points:Tonsil, eye and elbow.
  Interventions: Other: Placebo auricular acupressure

INTERVENTIONS:
Other: Auricular acupressure — The magnetic beads were taped to the auricular acupressure points, by the same acupuncture specialist on one ear approximately after skin sterilization, and the subjects were asked to massage the points for 5 minutes, 30 minutes before three meals and sleep.The magnetic beads were left in situ, but replaced with new ones once every week in the other ear.
  Arms: Auricular acupressure
Other: Placebo auricular acupressure — The magnetic beads were taped to the auricular acupressure points, by the same acupuncture specialist on one ear approximately after skin sterilization, and the subjects were not asked to massage the points.The magnetic beads were left in situ, but replaced with new ones once every week in the other ear.
  Arms: Placebo auricular acupressure

SUMMARY:
The purpose of this trial is to investigate the effect and safety of auricular acupressure on adolescent and young women with PCOS. Subjects will be randomly assigned in to two arms: Auricular acupressure arm and placebo auricular acupressure, both arms will be treated for three months. Body mass index, oral glucose tolerance test, hormonal profile and metabolic profile will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 12 and 25 years.
* Diagnosis of PCOS according to the modified Rotterdam criteria.
* 2 years after menarche.
* Body mass index (BMI) equal to or greater than 23 kg/m*m.

Exclusion Criteria:

* Administration of other medications known to affect reproductive function or metabolism within the past three months, including oral contraceptives, Gonadotropin-releasing hormone (GnRH) agonists and antagonists, anti androgens, gonadotropins, anti-obesity drugs, Chinese herbal medicines, anti diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, and calcium channel blockers.
* Patients with other endocrine disorders including 21-hydroxylase deficiency, hyperprolactinemia, uncorrected thyroid disease, suspected Cushing's syndrome.
* Patients with known severe organ dysfunction or mental illness.

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI): BMI change at 3 months. | 3 month

SECONDARY OUTCOMES:
Oral glucose tolerance test (OGTT) | 3 month
Testosterone (T) | 3 month
Sex hormone-binding globulin (SHBG) | 3 month
Dehydroepiandrosterone sulfate (DHEAS). | 3 month
Follicle stimulating hormone (FSH) | 3 month
Luteinizing hormone (LH) | 3 month
Cholesterol | 3 month
Triglycerides (TG) | 3 month
Waist/hip ratio | 3 month
Ferriman-Gallwey score | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Lihui Hou, Bachelor, Study Chair — First Affiliated Hospital of Heilongjiang University Of Chinese
Locations (1):
- First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China